CLINICAL TRIAL: NCT05968534
Title: MOSAIC (MOthers' AdvocateS In the Community) for Pregnant Women and Mothers of Children Under 5 With Experience of Intimate Partner Violence: Open Trial
Brief Title: MOSAIC (MOthers' AdvocateS In the Community) for Pregnant Women and Mothers of Children Under 5 With Experience of Intimate Partner Violence (MOSAIC Plus) Open Trial
Acronym: MOSAIC Plus OT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Maji Debena, Assistant Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 361186
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Intimate Partner Violence; Depression; Posttraumatic Stress Symptom
Keywords: women; mothers; pregnant
MeSH Terms: conditions — Depression | interventions — Mosaicism

STUDY DESIGN:
Intervention Model Description: "Mother AdvocateS In the Community (MOSAIC) Plus" intervention to reduce depressive and PTSD symptoms and prevent additional IPV among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate IPT principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOSAIC Plus (Other): This is a single-arm open-trial to evaluate and refine the feasibility and acceptability of training and recruitment methods. Data from this phase will be used to refine and inform study procedures for the subsequent RCT.
  Interventions: Behavioral: MOSAIC Plus

INTERVENTIONS:
Behavioral: MOSAIC Plus — This is a single-arm study. Participants will receive the intervention is called "Mother AdvocateS In the Community (MOSAIC) Plus", an intervention to reduce depressive and PTSD symptoms and prevent additional intimate partner violence among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate interpersonal psychotherapy principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms.

SUMMARY:
The purpose of this R34 exploratory research proposal is to conduct formative work for a larger randomized controlled trial (RCT) evaluating the effectiveness of the "Mother AdvocateS In the Community (MOSAIC) Plus" intervention to reduce depressive and PTSD symptoms and prevent additional IPV among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate IPT principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms. The proposed open trial will enroll 15 pregnant women who report experience of IPV in the past 6 months, and who screen positive for elevated depressive and/or PTSD symptoms. The intervention lasts 6 months after enrollment.

DETAILED DESCRIPTION:
Violence against women is a global human rights concern and a significant public health challenge; 1 in 3 three women experience lifetime physical and/or sexual violence. As many as 5.3 million U.S. women report experiencing intimate partner violence (IPV; referring to sexual or physical violence by current or former partners) annually. Depression and posttraumatic stress disorder (PTSD) are the two most common mental health consequences of IPV. In turn, developing depressive and PTSD symptoms after experiencing IPV increases future risk of IPV3. IPV is also associated with chronic physical health problems and self-harm .

Motherhood and pregnancy increase the risk for prolonged exposure to physical, psychological and sexual IPV. With as many as 4% to 8% of pregnant women reporting IPV during pregnancy, IPV can start or worsen during the perinatal period. Previous and current experience of IPV is strongly associated with poor physical health, mental health and obstetric outcomes; leading to increased utilization of health services11 even after the IPV ends12. There are very few interventions that effectively reduce IPV among pregnant women and mothers with children under 5 who report IPV. One of them, Mother AdvocateS In the Community (MOSAIC) forms the basis of this proposal16. No existing intervention addresses the depressive and PTSD symptoms that often follow IPV, are associated with suffering and morbidity, and potentiate future IPV risk for pregnant women and mothers with children under 5 who report IPV. In fact, there are not any interventions for any group of women that effectively reduce both future IPV risk and common related mental health symptoms such as depression and PTSD. An integrated intervention that addresses elevated symptoms of maternal depression and PTSD while reducing subsequent IPV is needed.

MOSAIC is a non-professional intervention delivered by mentor mothers from the community to reduce IPV in pregnant women and mothers with children under 5. The intervention combines elements of mentoring and IPV-specific support provided by mentor mothers. MOSAIC was also tested in a fully-powered RCT for pregnant women and mothers with children under 5 in Australia and found to reduce subsequent IPV. However, it did not significantly improve depression, and PTSD symptoms were not evaluated. Given the suffering, morbidity, and additional risk of IPV conferred by depressive and PTSD symptoms, the proposed study will augment MOSAIC with principles of an evidence-based intervention to improve maternal mental health. Interpersonal psychotherapy (IPT) is the front-line treatment for maternal depression18 and has been found to reduce PTSD symptoms in the perinatal period19. IPT addresses maternal mental health by helping women increase their general social support systems and build communication skills and confidence to access needed resources and help. IPT can be effectively delivered by lay providers. This proposal will integrate IPT principles into MOSAIC to address both IPV and its mental health sequelae.

The purpose of this R34 exploratory research proposal is to conduct formative work for a larger randomized controlled trial (RCT) evaluating the effectiveness of the "Mother AdvocateS In the Community (MOSAIC) Plus" intervention to reduce depressive and PTSD symptoms and prevent additional IPV among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate IPT principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms. The proposed study will enroll pregnant women who report experience of IPV in the past 6 months, and who screen positive for elevated depressive and/or PTSD symptoms. The intervention lasts 9 months after enrollment. Women will be recruited from Obstetrics and Gynecological unit of the Hurley Medical Center and YWCA, Flint. The control condition will be the original MOSAIC intervention. Study assessments will take place at baseline, 3, 6 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and/or are mothers of children under 5
* Report IPV experiences in the past 6 months (as assessed by Composite Abuse Scale)
* Aged 18 or above,
* Have elevated depressive and/or PTSD symptoms as assessed by Patient Health Questionnaire (PHQ-9) with a cutoff point of ≥9, and/or the Davidson Trauma Scale (DTS) with a cut-off point of ≥40.

Exclusion Criteria:

* Cannot provide the name and contact information of at least two locator persons,
* Do not have access to any telephone,
* Cannot understand English well enough to understand the consent form or assessment instruments when they are read aloud

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | 9 months
  Number of clients reporting acceptability of the proposed recruitment methods, research design, intervention training methods, and of delivering the MOSAIC Plus and MOSAIC interventions by using End of Treatment Questionnaire. The questionnaire assesses rate of recruitment and retention of participants and dropouts and rates of completion.
Satisfaction with care | 9 months
  Number of clients reporting satisfaction with care through rate of recruitment, client retention and intervention completion as reported in the Client Satisfaction Questionnaire,
Quality of working relationship | 9 months
  Evaluate therapeutic alliance by using Working Alliance Inventory-Short Revised (WAI-SR)
Changes in depressive symptoms | baseline, 3, 6 and 9 months
  Number of participants reporting changes in depressive symptoms as assessed by Patient Health Questionnaire (PHQ-9). Scores range from 0-27. Higher scores indicate severity of depressive symptoms.
Changes in posttraumatic stress disorder symptoms | baseline, 3, 6 and 9 months
  Number of participants reporting changes in posttraumatic stress disorder symptoms by using Davidson Trauma Scale. Higher scores indicate severity of posttraumatic stress symptoms.

SECONDARY OUTCOMES:
Changes in intimate partner violence | baseline, 3, 6 and 9 months
  Number of participants reporting changes in subsequent intimate partner violence by using Composite Abuse Scale. Higher scores indicate severity of intimate partner violence.
Effectiveness obtaining resources | baseline, 3, 6 and 9 months
  Number of participants reporting changes in effectiveness in obtaining resources by using Effectiveness Obtaining Resources (EOR) scale. Higher scores indicate improved effectiveness in obtaining resources.
Perceived social support | baseline, 3, 6 and 9 months
  Number of participants reporting changes in perceived social support by using The RAND social support scale (Medical Outcome Study-Social Support Survey MOS-SS). Higher scores demonstrate strength of social support.
Functioning | baseline, 3, 6 and 9 months
  Number of participants reporting changes in mental health related disability as evaluated by WHO Disability Assessment schedule-12. Higher scores demonstrate severity of mental health related disability.
Self-care and self-worth | baseline, 3, 6 and 9 months
  Number of participants reporting changes in self-care and self-worth as evaluated by self-care and self-worth scale.
General health and wellbeing | baseline, 3, 6 and 9 months
  Number of participants reporting changes in general health and wellbeing as evaluated by the SF-36 scale. Scale ranges 0-100 and higher scores indicate better health and wellbeing.

OTHER OUTCOMES:
Provider Competencies | 6 and 9 months
  Number of participants reporting on competency of providers by using Competency Assessment Inventory (CAI).
Quality of working relationship-provider perspective | 3, 6 and 9 months
  Assess the quality of working relationship by using the provider perspective section of working alliance inventory. The scale has scores ranging from 5 to 20. Higher scores indicate a better therapeutic alliance.

CONTACTS AND LOCATIONS:
Locations (1):
- YWCA-Flint, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided